CLINICAL TRIAL: NCT02631083
Title: The Impact of a Low Glycaemic Index (GI) Diet on Daily Blood Glucose Profiles and Energy Flux in Male Chinese Adults.
Brief Title: The Influence of Glucose Flux on Fat Synthesis in a Whole Body Calorimeter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2014/00960
Record Dates: First submitted 2015-12-11; First posted 2015-12-15 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Type 2 Diabetes, Obesity, Prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Prediabetic State | interventions — Breakfast; Lunch; Snacks; Meals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breakfast, lunch, snack and dinner (high GI) (Experimental): Subjects will consume meals which are high glycemic index for breakfast (Honey stars cereal), lunch (glutinous rice meal) and snack (white bread and jam) in the whole body calorimeter. A take-away high glycemic index dinner will be provided.
  Interventions: Other: Breakfast, lunch, snack and dinner
- Breakfast, lunch, snack and dinner (low GI) (Experimental): Subjects will consume meals which are low glycemic index for breakfast (All bran cereal), lunch (basmati rice meal) and snack (multigrain bread and sugar-free jam) in the whole body calorimeter. A take-away low glycemic index dinner will be provided.
  Interventions: Other: Breakfast, lunch, snack and dinner

INTERVENTIONS:
Other: Breakfast, lunch, snack and dinner — These meals (cereal, rice and bread meals) will be tested in subjects for their glycaemic response (CGMS) and substrate utilization (calorimeter)

SUMMARY:
The study is carried out to find out the inclusion of high and low glycaemic index foods to daily meals and how they impact 24 hour blood glucose fluctuations and energy regulation.

DETAILED DESCRIPTION:
The GI is a method of classifying foods based on the food's ability to raise the blood glucose level. Low GI foods are recommended as they have a lower impact on blood glucose concentrations. The research sets out to determine the effect of GI on 24 hour blood glucose profiles and energy regulation in Asians. Healthy, normal-weight, Chinese males will be recruited. There will be two sessions (consisting of four days for each session) where they will consume either a high or low GI breakfast, lunch, snack (in the whole body calorimeter), and a high or low glycaemic index dinner at home. They will take part in two test sessions (each spanning over 3 days) with at least five days in between the two sessions. Their glycaemic response will be measured using a Continuous Glucose Monitoring System (CGMS) throughout the period, while substrate oxidation will be measured over 10 hours in the calorimeter (from breakfast, lunch and snack). This study specifically attempts to see how having high and low GI meals impact on blood glucose levels and energy regulation in Asians. The study is important in that it will be the first of its kind in the whole body calorimeter and enable us to compute the rate of fat synthesis and how it is modulated when subjects are fed a high GI diet (increased glucose excursions) and a low GI diet ( blunted glucose) over 24 hours in healthy Asians. Obesity and diabetes rates are increasing exponentially in Asian populations and Singapore is no exception. Devising ways and means to staunch the escalation is therefore a priority. The findings of the research will contribute towards the long-term objectives of developing Asian specific dietary guidelines for weight and glycaemic control. The study data will also be important for the provision of practical food-based advocacy for better weight and glycaemic control in Singaporeans.

ELIGIBILITY:
Inclusion Criteria:

* Chinese, male
* Age between 21-40 years
* Body mass index between 17 to 25 kg/m2
* Normal blood pressure (<140/80 Hgmm)
* Fasting blood glucose < 6 mmol/L

Exclusion Criteria:

* Having any metabolic diseases (such as diabetes, hypertension etc)
* On prescription medication
* Having glucose 6-phosphate dehydrogenase deficiency (G6PD)
* Partaking in sports at the competitive and/or endurance levels
* Allergic/intolerant to any of the test foods
* Intentionally restricting food intake
* Smoking

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Glycaemic response The blood glucose response to low and high GI test foods measured 2 hours post consumption using the Continuous Glucose Monitoring System (CGMS) | 2 hours post consumption
  The blood glucose response to low and high GI test foods measured 2 hours post consumption using the Continuous Glucose Monitoring System (CGMS)
  The blood glucose response to low and high GI test foods measured 2 hours post consumption using the Continuous Glucose Monitoring System (CGMS)
Daily blood glucose profile | 24 hours
  The daily total blood glucose response is measured for each low and high GI treatment as the area under the curve over 24 hours using CGMS for breakfast, lunch, snack and dinner.
Substrate oxidation | 2 hours post consumption
  The carbohydrate and fat oxidation (i.e Respiratory Quotient) after consumption of low and high GI test foods measured 2 hours post consumption using indirect calorimetry in a whole body calorimeter. This is done over 10 hours in the whole body calorimeter measured for breakfast, lunch and snack only

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Derived] Camps SG, Kaur B, Quek RYC, Henry CJ. Does the ingestion of a 24 hour low glycaemic index Asian mixed meal diet improve glycaemic response and promote fat oxidation? A controlled, randomized cross-over study. Nutr J. 2017 Jul 12;16(1):43. doi: 10.1186/s12937-017-0258-1. PMID 28701162